CLINICAL TRIAL: NCT04650815
Title: Community Dynamics of Malaria Transmission in Humans and Mosquitoes at the Area of Sabou, Burkina Faso
Brief Title: Malaria Transmission in Humans and Mosquitoes at the Area of Sabou, Burkina Faso
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000135; 000135-I
Record Dates: First submitted 2020-12-02; First posted 2020-12-03 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05-16

CONDITIONS: Malaria
Keywords: Assays; BLOOD SAMPLING; Parasites; Gametocyte; Infection; Natural History
MeSH Terms: conditions — Malaria; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 0.5 - 5 Years: Infants and Children up to age 5 years in the Sabou Health District
- 10 - 18 Years: Children ranging in age 10 to 18 years in the Sabou Health District
- 19 + Years: Adults ranging in ages 19 years to 65 years in the Sabou Health District
- 5 - 10 Years: Children ranging in age 5 years through 10 years in the Sabou Health District

SUMMARY:
Background:

Malaria is a disease that affects many people in Burkina Faso. It is caused by germs that are spread by mosquito bites. A vaccine that blocks the spread of malaria is important to get rid of the disease. To see if a vaccine works, researchers need to find out how many malaria infections are happening in the community.

Objective:

To learn how often people of all ages who live in Sabou, Burkina Faso, get malaria.

Eligibility:

Healthy people ages 6 months to 65 years who reside in Sabou in a household with adults and children.

Design:

Participants will be screened with questions about their health. They will have a physical exam.

Participants will be asked about any malaria symptoms they are having. They will be asked about the use of bed nets. Their vital signs, like blood pressure and temperature, will be measured.

They will have blood taken from their arm with a needle.

Participants who have a fever will have a malaria test. Those who test positive for malaria will be referred to the local health facility for treatment.

Participants will have monthly study visits. Blood will be taken from a finger.

Participants may be invited to take part in 2 mosquito feeding experiments. Mosquitos that do not carry malaria will bite their arm. And a small amount of blood will be fed to mosquitos in a laboratory.

Participants' homes will be examined for mosquitoes. Researchers will remove all mosquitoes they collect. Participants' homes will be sprayed with a chemical to kill mosquitoes and other insects.

Participation will last for 12 months.

DETAILED DESCRIPTION:
A vaccine that interrupts malaria transmission is critical to eradicate the disease, but improved assays are needed to measure the efficacy of vaccines. Transmission-blocking vaccines (TBVs) work by inducing antibodies in vaccines that inhibit parasite development in the mosquito interrupting transmission. Efficacy of vaccines may be estimated by in vitro membrane feeding assays using immune sera and laboratory mosquitoes, but qualified assays that measure transmission in the field are needed to assess transmission-blocking interventions in natura. Clinical trials of TBV have started elsewhere on the continent in Mali, and we expect to expand TBV studies here in Burkina Faso in the future. This protocol will use a longitudinal cohort to gather information on the rates of blood smear positive individuals by month, season and year at Sabou Health district area, Burkina Faso. Individuals in the villages will be approached first for participation, including permission to contact their household and neighbors of their compound for participation. Households will be identified using census data and individuals will be consented for participation. Malaria smears will be obtained at monthly visits, in conjunction with mosquito collections in/around village residences. Parasite rates in locally caught mosquitoes will be assessed longitudinally for differences by season and year.

A total of 600 volunteers from Sabou area will be enrolled. Participants aged 0.5-65 years will have monthly blood sampling and mosquito collection at their household. Participants will be followed for up to 1 year, to collect data that will guide the design of future community-based trials of TBV.

ELIGIBILITY:
* HOUSEHOLD INCLUSION CRITERIA:

In order to be included in the study, households must meet all of the following inclusion criteria:

* Household with at least 3 residents eligible for participation.
* Household with at least one compound member who is below 5 years of age whose parents or caretakers are willing to provide informed consent for the child to participate
* Household with at least one compound member aged 5-15 years whose parents or caretakers are willing to provide informed consent for the child to participate
* Household members willing to accommodate mosquito sampling in their compound, both indoors and outdoors.

SUBJECT INCLUSION CRITERIA:

* 0.5 to 65 years of age
* Known resident within the study area and planning to remain for the duration of the study
* Acceptance and signature of the written informed consent and the assent for children aged 12-19 years who are not otherwise emancipated

SUBJECT EXCLUSION CRITERIA:

* Major congenital defect diagnosed based on medical history and examination
* Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Current participation in malaria vaccine trials or participation in such trials in the last 2 years

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Up to 900 volunteers (ages 0.5 - 65 years) from Sabou Health District area will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 608 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Measurement of blood smear positive individuals by age over the course of one year. These estimates will be stratified by age brackets of transmission interest (0.5-5, 5-10, 10-18, 19+ years old) | one year
  Monthly rates of blood smear positive individuals by age over the course of one year

CONTACTS AND LOCATIONS:
Overall Officials: Patrick E Duffy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Burkina Faso (2):
  - CMAMK, Sabou
  - GRAS, Sabou

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data because collected data will be used to guide the design of future community-based trials of TBV.